CLINICAL TRIAL: NCT06265831
Title: The Effect of Face Hand Fan Application on Dyspnea and Quality of Life in COPD Patients
Brief Title: The Effect of Face Hand Fan Application on Dyspnea
Acronym: HandfanCOPD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Necmiye ÇÖMLEKÇİ, Research Assistant, PhD, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BU-FHS-NC-03
Record Dates: First submitted 2024-02-10; First posted 2024-02-20 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: COPD
Keywords: dyspnea; COPD; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Intervention Model Description: Parallel group: two groups, an intervention group and a control group, receiving complementary therapy.
Who Masked: Participant
Masking Description: Hospitalized patients with a diagnosis of COPD will be randomized into two groups. The intervention group will have a hand fan applied to the face and be monitored for a week, and the control group will receive routine care at the clinic. Investigators will evaluate outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand-fan application to the face (Experimental): At the first meeting of the hand-fan application to the face group, the Patient Identification Form, Vital Signs Form, Modified Borg Scale, and Saint George Respiratory Questionnaire Form will be filled out. Afterward, training will be given (accompanied by an academic advisor) on how to apply cold air to the face with a hand fan (3 times a day for 5 minutes) for dyspnea management. Additionally, patients will be given a hand-fan application brochure. The researchers will monitor the patient every day for a week (7 days), fill out the vital signs form, and the final test will be administered by the researchers on the 8th day.
  Interventions: Other: Hand-fan application to the face
- Standard care group (No Intervention): In the standard care group, the Patient Diagnosis Form, Vital Signs Form, Modified Borg Scale, and Saint George Respiratory Questionnaire Form will be filled in at the first interview. The clinic's routine care protocol will be applied to the patients in the control group, and the researchers will fill out a vital signs form every day for a week, and the patients will be followed up.

INTERVENTIONS:
Other: Hand-fan application to the face — Hand fan application is one of the applications recommended in managing dyspnea in evidence-based guidelines. Hand fan application effectively reduces shortness of breath by stimulating cold airflow to the 2nd and 3rd trigeminal nerve branches, mucosa, and skin.
  Arms: Hand-fan application to the face

SUMMARY:
Diagnosing and managing dyspnea in patients with COPD is very important. Although pharmacological and non-pharmacological methods are used in the management of dyspnea, it is recommended that pharmacological methods be supported by non-pharmacological methods. Hand fan application, which is one of the non-pharmacological methods used in dyspnea management, provides an increase in self-efficacy in patients in addition to the stimulation of cold air flow to the trigeminal nerve branches, mucosa and skin. Although there are studies reporting that applying cold air to the face with a hand fan is effective in reducing the severity of dyspnea in different patient groups, the number of studies examining the effectiveness of applying cold air to the face with a hand fan in patients with COPD is quite limited. This project was planned to determine the effect of applying cold air to the face with a fan on the severity of dyspnea and quality of life in COPD patients.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a chronic disease with a high incidence both in our country and around the world. Dyspnea is one of the common problems in COPD patients. Dyspnea is an important symptom that limits patients' physical mobility, causes psychological problems such as anxiety, depression, and panic, and negatively affects their quality of life. Therefore, it is very important to diagnose and manage dyspnea in patients with COPD. Although pharmacological and non-pharmacological methods are used in the management of dyspnea, it is recommended that pharmacological methods be supported by non-pharmacological methods. Hand fan application, which is one of the non-pharmacological methods used in dyspnea management, provides an increase in self-efficacy in patients in addition to the stimulation of cold airflow to the trigeminal nerve branches, mucosa, and skin. Although there are studies reporting that applying cold air to the face with a hand fan is effective in reducing the severity of dyspnea in different patient groups, the number of studies examining the effectiveness of applying cold air to the face with a hand fan in patients with COPD is quite limited. This project was planned to determine the effect of applying cold air to the face with a fan on the severity of dyspnea and quality of life in COPD patients.

Method: The research was planned as a randomized, controlled experimental design. The population of the research consists of patients treated with a diagnosis of COPD in Bartın State Hospital Chest Diseases Service. Considering the data obtained from a similar study, the sample was calculated as 64 patients in the intervention group and 64 patients in the control group, for a total of 128 patients. Data will be collected using the Descriptive Information Form, Vital Signs Form, Modified Borg Scale, and Saint George Respiratory Questionnaire.

Data will be collected by researchers through face-to-face interviews with COPD patients treated at Bartın State Hospital Chest Diseases Service. Patients receiving treatment with a diagnosis of COPD will be randomized into intervention and control groups. In the control group, the Patient Diagnosis Form, Vital Signs Form, Modified Borg Scale, and Saint George Respiratory Questionnaire Form will be filled in at the first interview. The clinic's routine care protocol will be applied to the patients in the control group, and the researchers will fill out a vital signs form every day for 7 days, and the patients will be followed up. At the first meeting of the intervention group, the Patient Identification Form, Vital Signs Form, Modified Borg Scale, and Saint George Respiratory Questionnaire Form will be filled out. Afterward, training will be given (accompanied by an academic advisor) on how to apply cold air to the face with a hand fan (3 times a day for 5 minutes) for dyspnea management. Additionally, patients will be given a hand-fan application brochure. The researchers will monitor the patient every day for a week (7 days), fill out the vital signs form, and the final test will be administered by the researchers on the 8th day.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with COPD at least 6 months ago,
* Being over 18 years of age,
* No open wounds on the face for any reason,
* Lung cancer, tuberculosis, asthma etc. absence of other respiratory system diseases,
* Not having a hearing or speech impairment,
* Not having a cognitive disability
* Volunteering to participate in the research.

Exclusion Criteria:

* Being diagnosed with COPD less than 6 months ago,
* Being under 18 years of age,
* Having an open wound on the face for any reason,
* Lung cancer, tuberculosis, asthma etc. Having other respiratory system diseases,
* Having hearing and speech impairment,
* Having a cognitive disability
* Not volunteering to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Modified Borg Scale | a week (seven days)
  The Modified Borg Scale was first developed to measure the effort expended during physical exercise. Later, MBS was revised in 1982 and became a scale consisting of 12 items that diagnose the severity of dyspnea according to its degree. As the points on the scale increase, the severity of dyspnea increases (0: None, 0.5: Very very mild, 1: Very mild, 2: Mild, 3: Moderate, 4: Somewhat severe, 5: Severe, 6: 7: Very severe, 8: ….., 9: Very very serious, 10: Maximum). Although MBS was first used to define the severity of exertional dyspnea, it is now also used to evaluate the severity of resting dyspnea.

SECONDARY OUTCOMES:
Saint George Respiratory Questionnaire | a week (seven days)
  Saint George Respiratory Questionnaire is a survey developed to evaluate the health-related quality of life of patients diagnosed with COPD. The survey consists of 50 items and 3 main sections. These sections; symptoms (8 items), activity (16 items) and effects of the disease (26 items). The questionnaire evaluates respiratory symptoms, activities restricted due to dyspnea, and the impact of this condition on daily life. In the evaluation, the total score of the survey is distributed between 0 and 100. A score of 0 indicates that there is no deterioration in the quality of life, while a score of 100 indicates that the quality of life is increasingly negatively affected. In the reliability analysis of SGSA, Cronbach's alpha coefficient was found to be 0.88 for the entire scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmiye ÇÖMLEKÇİ, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After the research is published as an article, the data will be shared with researchers who request it. (Personal and private information of the participants is hidden.)
Supporting Information: Study Protocol, SAP